CLINICAL TRIAL: NCT03908788
Title: Detection of the Emergence of RAS (Rat Sarcoma Viral Oncogene Homolog) Mutations in Circulating DNA (Deoxyribonucleic Acid) in Patients With Metastatic Colorectal Cancer During Treatment With Anti-EGFR (Epidermal Growth Factor Receptor) Therapy
Brief Title: Detection of the Emergence of RAS (Rat Sarcoma Viral Oncogene Homolog) Mutations in Circulating DNA (Deoxyribonucleic Acid) in Patients With mCRC (Metastatic Colorectal Cancer) During Treatment With Anti-EGFR (Epidermal Growth Factor Receptor) Therapy
Acronym: EmutRAS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-A00232-53
Record Dates: First submitted 2019-01-25; First posted 2019-04-09 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer; Detection of the emergence of RAS mutations; Circulating DNA in patients; Treatment with anti-EGFR therapy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intplex test (Experimental): In vitro diagnostic device
  Interventions: Device: Intplex test

INTERVENTIONS:
Device: Intplex test — Blood sample at each tumor assessment

SUMMARY:
The analysis of circulating DNA (Deoxyribonucleic acid) to identify potential resistance mechanisms during anti-EGFR (epidermal growth factor receptor) treatment is of great interest, as evidenced by the recent journal published by Corcoran in the prestigious New England Journal of Medicine.

EmutRAS is one of the first studies that will specifically and prospectively evaluate the RAS mutational switch and its impact on the efficiency of the 1st line processing.

DETAILED DESCRIPTION:
The primary study objective is the Detection of RAS mutational (rat sarcoma viral oncogene homolog) "switch" in circulating DNA by Intplex® test in mCRC (metastatic colorectal cancer) patients treated with antibody anti-EGFR (epidermal growth factor receptor), cetuximab or panitumumab in first line.

The treatment and these modalities will be decided by the investigator.

The study is based on blood sampling, the frequency of which is described below, rhythm of plasma samples:

Inclusion after determination of wild status RAS tissues.

First sampling of 2 EDTA (ethylenediaminetetraacetic acid) tubes, then at each tumour evaluation during treatment with anti EGFR (epidermal growth facor receptor), every 4 cures. At the end of treatment or after more than 36 treatment cures, a final sample will be taken.

No results of the samples will be communicated to the investigator, the sponsor will centralize these results for the final analysis of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically confirmed metastatic colorectal cancer
* Patient treated in the first line by one of the treatments below and according to a bi-monthly schema for cetuximab: FOLFIRI (elvorin + 5 Fluorouracil + irinotecan) ou FOLFOX (elvorin + 5 Fluorouracil + oxalplatin) + Cetuximab* (Erbitux) ; FOLFIRI ou FOLFOX + Panitumumab (Vectibix); FOLFIRINOX ou FOLFOXIRI ((elvorin + 5 Fluorouracil + oxaliplatin + irinotecan) + Cetuximab* (Erbitux); FOLFIRINOX ou FOLFOXIRI + Panitumumab (Vectibix) For patient treated cetuximab administration will be bi-monthly
* Patient with at least one evaluable metastatic target according to RECIST 1.1 (Response Evaluation Criteria in Solid Tumors)
* Wild RAS (rat sarcoma viral oncogene homolog) status detected by standard tissue test, on primary tumor and / or metastasis
* Wild BRAF (murine sarcoma viral oncogene homolog B) status detected by standard tissue test, on primary tumor and / or metastasis
* Man or woman> 18 years old
* Signed informed consent before any specific procedure to study
* Patient affiliated to the social security or equivalent

Exclusion Criteria:

* Previous treatment with an anti-EGFR (epidermal growth factor receptor)
* Patient with a multifocal primary tumor
* RAS (rat sarcoma viral oncogene homolog) status mutated or not detectable on tissue analysis
* BRAF (murine sarcoma viral oncogene homolog B) status mutated or undetectable on tissue analysis
* Patient receiving adjuvant chemotherapy or radiotherapy within <14 days
* History of other cancer in the last 5 years (except in-situ carcinoma of the cervix and cutaneous carcinoma excluding melanoma treated optimally)
* Blood transfusion (whole blood, red blood cell, platelets...) in the previous week
* Patients with psychological, familial, sociological or geographic conditions potentially not favorable to the good observance of the study protocol and the follow-up
* Legal incapacity or limited legal capacity

Participation in another interventional clinical trial - biomedical research (therapeutic strategy type) is not excluded provided that it is use an Anti-EGFR with a AMM (marketing authorization), (Cetuximab - Panitumumab) with a dose and a standard administration rhythm (according to the AMM).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2018-07-26 (Actual); Primary Completion 2023-12-03 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with mCRC (metastatic colorectal cancer) who develop a RAS (rat sarcoma viral oncogene homolog) mutation under anti-EGFR (epidermal growth factor receptor) therapy | Approximately 8 weeks
  From baseline to the end of treatment

SECONDARY OUTCOMES:
Probability of obtaining a positive test, i.e. RAS status mutated by the Intplex® test, among the patients determined RAS mutated by the tissue test | Approximately 8 weeks
  From baseline to the end of treatment
Probability of obtaining a negative test, i.e. wild RAS status by the Intplex® test among patients determined wild RAS by the tissue test | Approximately 8 weeks
  From baseline to the end of treatment
Probability of obtaining a positive test, i.e. BRAF status mutated by the Intplex® test, among the patients determined BRAF mutated by the tissue test | Approximately 8 weeks
  From baseline to the end of treatment
Probability of obtaining a negative test, i.e. wild BRAF status by Intplex® test among patients determined wild BRAF by tissue test.compared to the pre-treatment tissue test | Approximately 8 weeks
  From baseline to the end of treatment
Proportion of patients with a BRAF mutation under anti-EGFR therapy | Approximately 8 weeks
  From baseline to the end of treatment
Progression-free survival | Approximately 36 months
  From baseline to the database cutoff
Global survival | Approximately 36 months
  From baseline to the database cutoff
Evaluation of the following criterion: total concentration of circulating DNA | Approximately 8 weeks
  From baseline to the end of treatment
Evaluation of the following criterion: integrity index | Approximately 8 weeks
  From baseline to the end of treatment
Evaluation of the following criterion: concentration of mutated alleles | Approximately 8 weeks
  From baseline to the end of treatment
Evaluation of the following criterion: frequency of mutated alleles | Approximately 8 weeks
  From baseline to the end of treatment

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - ICM Val d'Aurelle, Montpellier, Montpellier
  - Institut du Cancer de Montpellier - Val d'Aurelle, Montpellier

IPD SHARING:
Plan to Share IPD: No